CLINICAL TRIAL: NCT00509821
Title: Enzastaurin Before and Concomitant With Radiation Therapy, Followed by Enzastaurin Maintenance Therapy in Patients With Newly Diagnosed Glioblastoma Without Methylation of the Promoter Gene of MGMT Enzyme - a Phase II Study
Brief Title: Enzastaurin Before and Concomitant With Radiation, Followed by Enzastaurin in Participants With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11491; H6Q-MC-S039 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-01

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — enzastaurin; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enzastaurin Once Daily (QD) (Experimental): Enzastaurin given orally (PO) once daily (QD). 1125 mg loading dose D(-)7 then 500 mg PO,QD with concomitant radiotherapy.
  Interventions: Drug: Enzastaurin 500 milligram (mg) Once Daily (QD)
- Enzastaurin Twice Daily (BID) (Experimental): Enzastaurin 1125 mg loading dose D(-)7 then 250 mg twice daily (BID) PO, with concomitant radiotherapy.
  Interventions: Drug: Enzastaurin 250 mg Twice Daily (BID)

INTERVENTIONS:
Drug: Enzastaurin 500 milligram (mg) Once Daily (QD) — 1125 mg loading dose D(-)7 then 500 mg QD, oral, daily until disease progression, given with and without radiotherapy treatment.
  Other Names: LY317615
  Arms: Enzastaurin Once Daily (QD)
Drug: Enzastaurin 250 mg Twice Daily (BID) — 1125 mg loading dose D(-)7 then 250 mg BID, oral, daily until disease progression, given with and without radiotherapy treatment.
  Other Names: LY317615
  Arms: Enzastaurin Twice Daily (BID)

SUMMARY:
The purpose of the protocol was to induce a novel radiochemotherapy with enzastaurin as first-line treatment regimen in glioblastoma: Participants with active, unmethylated MGMT promoter were treated with enzastaurin before, concomitant, and after radiotherapy to determine safety and PFS at 6 months (PFS-6) in phase II.

ELIGIBILITY:
Inclusion Criteria:

* Present with newly diagnosed histologically proven supratentorial GBM.
* Demonstration of an unmethylated MGMT-promotor
* Participants must sign an informed consent document. Participants must be at least 18 years of age.
* Estimated life expectancy of at least 12 weeks
* Tumor tissue specimens (paraffin-embedded and/or frozen) from the GBM surgery or biopsy must be available for central pathology review and exploratory analysis of PKC-beta targets (for example, GSK3beta).
* Disease evaluated by Gd-MRI (magnetic resonance imaging) within 72 hours postoperatively
* Interval of greater than or equal to 2 and less than or equal to 4 weeks since surgery or biopsy
* ECOG Performance Status of less than or equal to 2
* Adequate organ function including the following:
* adequate bone marrow reserve: white blood cell (WBC) count greater than or equal to 3.0 X 109/L, absolute neutrophil count (ANC) greater than or equal to 1.5 X 109/L, platelet count greater than or equal to 75.0 X 109/L, and hemoglobin greater than or equal to 10.0 g/dL (greater than or equal to 6.2 mmol/L).
* Hepatic: bilirubin less than or equal to 1.5 times the upper limit of normal (X ULN), alkaline phosphatase (ALP), aspartate transaminase (AST), and alanine transaminase (ALT) less than or equal to 2.5 X ULN, or less than or equal to 5 X ULN with liver metastases
* Renal: serum creatinine less than or equal to 1.5 X ULN
* Blood clotting: prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits
* Participants must discontinue use of enzyme-inducing antiepileptic drugs (EIAEDs) greater than or equal to 14 days prior to study enrollment. The investigator may prescribe non-EIAEDs. Participants who must begin EIAED therapy while on study will be allowed to remain on study.
* Clinically normal cardiac function without history of ischemic heart disease in the past 6 months and normal 12-lead electrocardiogram (ECG); no history of stroke

Exclusion Criteria:

* Have a prior malignancy (other than glioblastoma, or adequately treated carcinoma in situ of the cervix, or nonmelanoma skin cancer), unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence
* Unable to undergo Gd MRI
* Prior chemotherapy within the last 5 years
* Prior chemotherapy for a brain tumor
* Prior radiotherapy of the head
* Are unable to discontinue use of carbamazepine, phenobarbital, and phenytoin
* History of coagulation disorder associated with bleeding, or recurrent thrombotic events
* Are receiving concurrent administration of anticoagulant therapy
* Placement of Gliadel® wafer at surgery
* Have a serious concomitant systemic disorder (for example, active infection including HIV, or cardiac disease) - participants who are pregnant, anticipate becoming pregnant within 6 months after study participation, or are currently breast-feeding
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- Germany (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regensburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers were defined as participants who had failure event(progressive disease, death), or were off treatment or censored due to study completion. Participants completed follow-up after receiving 1 dose of study drug and a post dose efficacy evaluation.
Groups:
- Enzastaurin Once Daily (QD): A loading dose of 1125 mg of enzastaurin administered orally (PO) on Day -7 (3 tablets of 125 mg, given 3 times daily (TID) followed by 500 mg once daily (QD)
- Enzastaurin Twice Daily (BID): A loading dose of 1125 mg of enzastaurin administered PO Day -7 (TID); the dose from Day -6 until study end was 500 mg, given in 2 daily PO (BID) doses of 250 mg
Period: Study Period 1 (Induction)
Arm/Group | Enzastaurin Once Daily (QD) | Enzastaurin Twice Daily (BID)
Started | 3 | 57
Received at Least 1 Dose of Study Drug | 3 | 57
Completed | 3 | 53
Not Completed | 0 | 4
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Progressive Disease | 0 | 1
Period: Study Period 2 (Radiation)
Arm/Group | Enzastaurin Once Daily (QD) | Enzastaurin Twice Daily (BID)
Started | 3 (Participants moved to Radiation Phase.) | 53 (Participants moved to Radiation Phase.)
Completed | 3 | 0
Not Completed | 0 | 53
Period: Study Period 3 (Maintenance)
Arm/Group | Enzastaurin Once Daily (QD) | Enzastaurin Twice Daily (BID)
Started | 3 | 49 (4 participants completed Radiation Phase but did not enter Maintenance Phase.)
Completed | 3 | 0
Not Completed | 0 | 49
Period: Study Period 4 (Follow Up)
Arm/Group | Enzastaurin Once Daily (QD) | Enzastaurin Twice Daily (BID)
Started | 2 (1 Participant completed Maintenance Phase but did not enter Follow-Up.) | 50 (1 Participant completed Radiation Phase, did not enter Maintenance Phase but entered Follow Up.)
Completed | 2 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enzastaurin QD participants data not collected, as per protocol. Enzastaurin BID are participants who received at least one dose of drug.
Groups:
- Enzastaurin Twice Daily (BID): Enzastaurin 1125 mg loading dose D(-)7 then 250 mg twice daily (BID) PO.
- Total: Total of all reporting groups
Arm/Group | Enzastaurin Once Daily (QD) | Enzastaurin Twice Daily (BID) | Total
Number analyzed (Participants) | 0 | 57 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data not collected as per protocol.
  years |  | 55.6 (11.29) | 55.6 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not collected as per protocol.
  Participants
    Female |  | 21 | 21
    Male |  | 36 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected as per protocol.
  Participants
    Hispanic or Latino |  | 57 | 57
    Not Hispanic or Latino |  | 0 | 0
    Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected as per protocol.
  Participants
    American Indian or Alaska Native |  | 0 | 0
    Asian |  | 0 | 0
    Native Hawaiian or Other Pacific Islander |  | 0 | 0
    Black or African American |  | 0 | 0
    White |  | 57 | 57
    More than one race |  | 0 | 0
    Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 0 | 57 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival at 6 Months (PFS-6)
Description: PFS-6 is defined as the percentage of participants with PFS at 6 months from the date of diagnosis to the first date of objectively determined progressive disease (based on radiological assessment) or death from any cause. It is assumed that PFS follows an exponential distribution.Estimation using Kaplan-Meier technique.
Time Frame: Baseline to 6 months
Population: All participants in BID arm who received at least one dose of study drug, BID, 4 participants were censored. Enzastaurin QD participants data not collected, as per protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin Twice Daily (BID)
Number analyzed (Participants) | 57
percentage of participants | 53.6 [39.8 to 65.6]

2. Secondary Outcome: Percentage of Participants With Overall Survival at 1 and 2 Years After Surgery
Description: Overall survival (OS) time is defined as the time from the date of diagnosis to the date of death from any cause. For participants who are still alive at the time of analysis, survival time will be censored at the last contact date. OS rate at 1 year (respectively 2 years) is determined using the OS times.
Time Frame: Baseline to 1 and 2 year
Population: All participants in BID arm who received at least one dose of study drug, BID, 11 participants were censored. Enzastaurin QD participants data not collected, as per protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin Twice Daily (BID)
Number analyzed (Participants) | 57
percentage of participants
  1 year | 63.0 [49.1 to 74.1]
  2 year | 27.0 [16.2 to 39.0]

3. Secondary Outcome: Response Rate
Description: Response rate is calculated as the number of participants with best response: complete response(CR: disappearance of all enhancing tumor on consecutive CT or magnetic resonance imaging (MRI) scans at least 1 month apart, off steroids, and neurologically stable or improved ) or partial response (PR:-50% reduction in size of enhancing tumor on consecutive CT or MRI scans at least 1 month apart, steroids stable or reduced, and neurologically stable or improved), divided by the number of participants treated, multiplied by 100. CR and PR were assessed according to the criteria defined by MacDonald et al. 1990. A CR or PR must be confirmed by a second assessment, performed ≥28 days after the first evidence of response.
Time Frame: Baseline to 30 months
Population: All participants in BID arm who received at least 1 dose of study drug. Enzastaurin QD participants data not collected, as per protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin Twice Daily (BID)
Number analyzed (Participants) | 57
percentage of participants | 7.0 [2.0 to 17.0]

4. Secondary Outcome: Change in Neurologic Status as Measured by Mini Mental Status Questionnaire, Total Score
Description: Mini Mental State Status questionnaire is 11 questions, total score can range from 0 to 30, with a higher score indicating better function and a negative change in baseline indicating decrease in cognitive function.
Time Frame: Baseline through Week 12 .
Population: All participants in BID arm who received at least 1 dose of study drug and had evaluable data. Enzastaurin QD participants data not collected, as per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzastaurin Twice Daily (BID)
Number analyzed (Participants) | 56
units on a scale | 28.3 (4.86)

ADVERSE EVENTS:
Time Frame: First dose of study drug through 4 years.
Description: All participants who received at least 1 dose of enzastaurin, Follow-up was included in Entire Study Arm.
Groups:
- Induction Enzastaurin Once Daily (QD): A loading dose of 1125 mg of enzastaurin administered orally (PO) on Day -7 (3 tablets of 125 mg, given 3 times daily (TID) followed by 500 mg once daily (QD)
- Induction Enzastaurin Twice Daily (BID): A loading dose of 1125 mg of enzastaurin administered PO Day -7 (TID); the dose from Day -6 until study end was 500 mg, given in 2 daily PO (BID) doses of 250 mg
- Radiation Enzastaurin Once Daily (QD): Enzastaurin 500 mg administered PO QD.
- Radiation Enzastaurin Twice Daily (BID): Enzastaurin 500 mg administered PO BID.
- Maintenance Enzastaurin Once Daily (QD): Enzastaurin 500 mg administered PO, QD continued until progression or unacceptable adverse events (AEs)
- Maintenance Enzastaurin Twice Daily (BID): Enzastaurin 500 mg administered PO, BID continued until progression or unacceptable adverse events (AEs)
- Enzastaurin Once Daily (QD) Entire Study; Enzastaurin Twice Daily (BID) Entire Study: A safety follow-up performed after end of enzastaurin treatment for all participants who received at least 1 dose of study drug.
Arm/Group | Induction Enzastaurin Once Daily (QD) | Induction Enzastaurin Twice Daily (BID) | Radiation Enzastaurin Once Daily (QD) | Radiation Enzastaurin Twice Daily (BID) | Maintenance Enzastaurin Once Daily (QD) | Maintenance Enzastaurin Twice Daily (BID) | Enzastaurin Once Daily (QD) Entire Study | Enzastaurin Twice Daily (BID) Entire Study
Serious Adverse Events (participants affected / at risk) | 0/3 | 5/57 | 0/3 | 16/53 | 0/3 | 8/49 | 0/3 | 27/57
Other Adverse Events (participants affected / at risk) | 3/3 | 22/57 | 3/3 | 43/53 | 3/3 | 28/49 | 3/3 | 50/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Enzastaurin Once Daily (QD) (N=3) | Induction Enzastaurin Twice Daily (BID) (N=57) | Radiation Enzastaurin Once Daily (QD) (N=3) | Radiation Enzastaurin Twice Daily (BID) (N=53) | Maintenance Enzastaurin Once Daily (QD) (N=3) | Maintenance Enzastaurin Twice Daily (BID) (N=49) | Enzastaurin Once Daily (QD) Entire Study (N=3) | Enzastaurin Twice Daily (BID) Entire Study (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (7) | 0 (0) | 6 (9)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Enzastaurin Once Daily (QD) (N=3) | Induction Enzastaurin Twice Daily (BID) (N=57) | Radiation Enzastaurin Once Daily (QD) (N=3) | Radiation Enzastaurin Twice Daily (BID) (N=53) | Maintenance Enzastaurin Once Daily (QD) (N=3) | Maintenance Enzastaurin Twice Daily (BID) (N=49) | Enzastaurin Once Daily (QD) Entire Study (N=3) | Enzastaurin Twice Daily (BID) Entire Study (N=57)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 7 (9)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 8 (8)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 4 (4) | 1 (1) | 9 (11)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (7) | 0 (0) | 9 (9)
Fatigue (General disorders) | 0 (0) | 4 (4) | 0 (0) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 13 (13)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 3 (5)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (10) | 3 (3) | 6 (13)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 3 (4)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (6)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 4 (5)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 6 (7)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 10 (12) | 0 (0) | 3 (3) | 2 (2) | 14 (20)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 9 (9)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 3 (3) | 9 (9) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 12 (12) | 0 (0) | 1 (1) | 3 (3) | 13 (13)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
3 participants receiving 500 mg enzastaurin qd were not included in analysis for outcome measures per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days